CLINICAL TRIAL: NCT01035437
Title: A Pilot Study for Determination of Feasibility and Toxicity of Pre-Treatment With HPPH (2-1[1-Hexyloxyethyl]-2 Devinyl Pyropheophorbide-a) Photodynamic Therapy Prior to Chemoradiation in Non-Operable Patients With Obstructive Esophageal Cancer
Brief Title: Study for Determination of Feasibility and Toxicity of Pre-Treatment With HPPH (2-1[1-Hexyloxyethyl]-2 Devinyl Pyropheophorbide-a) Photodynamic Therapy Prior to Chemoradiation in Non-Operable Patients With Obstructive Esophageal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPCI I 148809
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Esophageal Neoplasm
Keywords: obstructing
MeSH Terms: conditions — Esophageal Neoplasms | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPPH (Experimental): HPPH
  Interventions: Drug: HPPH 2-1[1-hexyloxyethyl]-2-devinyl Pyropheophorbide-a)

INTERVENTIONS:
Drug: HPPH 2-1[1-hexyloxyethyl]-2-devinyl Pyropheophorbide-a) — HPPH in D5W, 4.0 mg/m2 infused over 1 hour

SUMMARY:
This study aim is to find out what effects capecitabine, oxaliplatin and radiation therapy following photodynamic therapy have on esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Partially or completely obstructing primary esophageal carcinoma, clinical stage I-IVa as determined by endoscopy, CT-scan, PET +/- endoscopic ultrasound. For distal esophagus tumors involving the GE junction, at least 50% or greater of the tumor bulk should be in the distal esophagus
* Ineligible for or refused surgical resection
* No Prior therapy allowed for esophageal cancer
* ECOG Performance status 0-1
* Life expectancy > 4 months
* Adequate hematologic parameters (hemoglobin> 9g/dl, ANC > 1500/ul, Platelets > 100,000/ul)
* Adequate biochemical parameters (total bilirubin and creatinine within institutional limits, AST and alkaline phosphatase less tham or equal to 3xUNL)
* Age > 18 years
* Signed informed consent
* Bronchoscopy with biopsy and cytology if primary esophageal cancer is < 26 cm from incisors
* Female patients of childbearing potential should have a negative serum or urine pregnancy test within 7 days prior to registration
* Patients of Childbearing potential agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method
* Both men and women and members of all races and ethnic are eligible for this trial

Exclusion Criteria:

* Hypersensitivity to platinum compounds, fluoropyrimidines or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this trail
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements
* Peripheral neuropathy ≥ Grade 2
* History of second malignancy within the previous years except for curatively treated carcinoma of the cervix in-situ or non-melanomatous skin cancer
* Patients who are pregnant or lactating
* Porphyria or hypersensitivity to porphyrin-like compounds
* Patients with known HIV or Hepatitis B or C (active, previously treated or both)
* Patients with tracheal or bronchial involvement, as determined by bronchoscopy
* Patients with documented unilateral or bilateral vocal cord paralysis
* Patients with T4 lesions by CT, MRI or EUS involving the aorta, lung or pericardium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Determine the toxicity of sequential PDT and chemoradiation in obstructing esophageal cancer | 2 year

SECONDARY OUTCOMES:
Evaluate the efficacy of PDT in palliation of dysphagia | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, MD, Principal Investigator — Roswell Park Cancer Institute